CLINICAL TRIAL: NCT01539252
Title: Examining the Impact of Using Two Dialysers in Parallel on Dialysis Adequacy in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Marcello Tonelli, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DDphos1
Record Dates: First submitted 2012-02-03; First posted 2012-02-27 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; adequacy; phosphate clearance; double dialyzer; two dialyzers in parallel
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dialyzer (Active Comparator): Single dialyzer
  Interventions: Procedure: Single dialyzer
- Double dialyzer (Experimental): Two dialyzers in parallel
  Interventions: Procedure: Two dialyzers

INTERVENTIONS:
Procedure: Single dialyzer — Hemodialysis treatment using a single Baxter dialyzer - considered standard hemodialysis treatment.
  Arms: Single dialyzer
Procedure: Two dialyzers — Hemodialysis treatment using a two Baxter dialyzers in parallel.
  Arms: Double dialyzer

SUMMARY:
The purpose of this study is to investigate the effectiveness of using two dialysers to lower the blood mineral levels in people receiving hemodialysis as compared to using one dialyser (usual treatment).

DETAILED DESCRIPTION:
Higher levels of serum phosphate are independently associated with an increased risk of death in hemodialysis patients. Therefore, there has been considerable interest in controlling serum phosphate while minimizing oral calcium load. While most attention has focused on the use of non-calcium containing phosphate binders such as sevelamer and lanthanum, modifying conventional dialysis regimens to improve phosphate clearance is an alternative approach that remains relatively unstudied. A secondary analysis of a previous randomized cross-over study from our group found that the use of two dialysers in parallel resulted in a reduction in pre-dialysis serum phosphate levels. As this study was small, and the mechanisms resulting in the reduction in phosphate levels were unclear, further study is warranted. The investigators will conduct a randomized cross-over study comparing the impact of dialyzing using two dialysers in parallel with a single dialyser in hyperphosphatemic hemodialysis patients.

There will be a total of 34 participants from Alberta,Canada participating in this study. The length of study participation is 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients must be on a stable regimen of hemodialysis for ≥ 3 months ('stable' defined as not expected to require a change to the duration or frequency of treatments)
* Serum phosphate > 1.6 mmol/l on last two consecutive lab tests at least 3 weeks apart (KDOQI guidelines recommend maintaining predialysis phosphate < 1.8mmol/l - as such, phosphate lowering in this subgroup of patients is particularly relevant)
* Patients must be on stable doses of a phosphate binder with no changes in dose 1 month prior to study enrolment.
* Blood flow rate ≥ 350 ml/min through a well-functioning access (This will exclude patients receiving inadequate dialysis due to a temporary venous dialysis catheter and will ensure sufficient blood flow to permit dialysis using two dialysers in parallel.)

Exclusion Criteria:

* Patients who have a scheduled renal transplant, change in dialysis modality, surgery or hospitalization or plan on moving away from the study site in the next three months.
* Patients with a projected life expectancy of less than 3 months.
* Patients with a contraindication to intra-dialytic anticoagulation. (Some patients require a small increase in the amount of anticoagulation required to prevent dialyser clotting when using two dialysers in parallel).
* Patients who have missed >8 dialysis treatments in the past 3 months.
* Patients with a dialysis regimen of >3 runs per week.
* Failure to provide informed consent.
* Patients enrolled in another (interventional) trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dialysate clearance of phosphate | 3 weeks
  Dialysate phosphate clearance levels in double dialyzer periods compared to single dialyzer periods.

SECONDARY OUTCOMES:
Serum phosphate | 3 weeks
  Serum phosphate levels in the double dialyzer periods compared to the single dialyzer periods.
Dialysate removal of phosphate | 3 weeks
  Dialysate removal levels of phosphate in the double dialyzer periods compared to the single dialyzer periods.

OTHER OUTCOMES:
Proportion of participants with serious adverse events | 30 days following last day of intervention
  The proportion of participants during the double dialyzer period compared to the single dialyzer period experiencing serious adverse events resulting in death, life threatening illness, hospitalization or prolongation of existing hospitalization, or persistent or significant disability.
Proportion of participants with adverse events | 30 days following last day of intervention
  The proportion of participants with adverse events (and by each type of adverse event) during the double dialyzer intervention compared to single dialyzer intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Tonelli, MD, Principal Investigator — University of Alberta; Braden Manns, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thompson S, Manns B, Lloyd A, Hemmelgarn B, MacRae J, Klarenbach S, Unsworth L, Courtney M, Tonelli M. Impact of using two dialyzers in parallel on phosphate clearance in hemodialysis patients: a randomized trial. Nephrol Dial Transplant. 2017 May 1;32(5):855-861. doi: 10.1093/ndt/gfw085. PMID 27190374